CLINICAL TRIAL: NCT02991690
Title: Systemic Hypothermia in Acute Cervical Spinal Cord Injury - A Prospective, Multi-center Case Controlled Study
Brief Title: Systemic Hypothermia in Acute Cervical Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Allan D. Levi, Professor and Chairman of Neurological Surgery, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160758; CDMRP-SC150063 (Other Grant/Funding Number: United States Department of Defense); 20160365 (Other: University of Miami IRB)
Record Dates: First submitted 2016-12-07; First posted 2016-12-13 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury, Acute
Keywords: Hypothermia; Cervical Spinal Cord Injury; Trauma
MeSH Terms: conditions — Spinal Cord Injuries; Hypothermia; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypothermia (Experimental): Intravascular hypothermia will be initiated within 24 hours post-injury and 33 degrees Celsius will be maintained for 48 hours.
  Interventions: Other: Hypothermia
- Control (No Intervention): Standard of care medical treatment, specific to each individual.

INTERVENTIONS:
Other: Hypothermia — To deliver intravascular hypothermia, an Alsius Icy CoolGuard® catheter (US Food and Drug Administration approved, Premarket Notification [510(k), K030421]; Alsius Corporation, Irvine, California) will be inserted through the femoral vein using a sterile technique. Patients will be cooled at a maximum rate (2-2.5 ºC/hr.) until they reach the target temperature (T 33 ºC), which will be maintained for 48 hours, and then re-warmed at 0.1 ºC/hr. until normothermia (T 37ºC) is achieved.
  Arms: Hypothermia

SUMMARY:
This study is a prospective multi-center trial designed to determine the safety profile and efficacy of modest (33ºC) intravascular hypothermia following acute cervical (C1 to C8) Spinal Cord Injury (SCI).

DETAILED DESCRIPTION:
The purpose of the proposed clinical trial is to demonstrate the safety and efficacy of intravascular hypothermia as part of the early hospital management and treatment for acute cervical SCI. Each year in the US, there are over 11,000 new cases of para- and quadriplegia and 100,000 new cases of partial but permanent neurological losses due to acute SCI. Thus the potential for clinical hypothermia following SCI to improve neurological outcome has significant value. Many patients suffering SCI become permanently dependent on caretakers and become a financial liability to both the family and society. Hypothermia has the potential to improve outcome so that more patients suffering SCI can regain independent motor and sensory function and remain economically productive members of society. The use of modest hypothermia through intravascular cooling may ultimately lead to better care of the patient with acute SCI and may also have more widespread uses in patients presenting with stroke or cardiac arrest. In the long-term, this research may lend support to the use of hypothermia that could in turn save money for the patients, hospitals, the government and society as a whole.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 70 years of age
* AIS Grade A - C
* Glasgow Coma Scale ≥14
* Able to start hypothermia treatment within 24 hours of injury
* Non-penetrating injury. Patients urgently taken to the operating room for surgical reduction may also be included.

Exclusion Criteria:

* Age > 70 years
* AIS Grade D
* Hyperthermia on admission (>38.5ºC)
* Severe systemic injury
* Severe bleeding
* Pregnancy
* Coagulopathy
* Thrombocytopenia
* Known prior severe cardiac history
* Blood dyscrasia
* Pancreatitis
* Reynaud's syndrome
* Cord transection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-08-04 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Neurological improvement on American Spinal Injury Association (ASIA) | Between baseline and 12 months
  Improvement in ASIA Impairment Scale (AIS) after modest hypothermia
Neurological improvement on ASIA | Between baseline and 12 months
  Improvement in ASIA motor score after modest hypothermia

SECONDARY OUTCOMES:
Functional improvement in Functional Independence Measure (FIM) | 12 months
  Functional improvement in FIM after modest hypothermia
Functional improvement in Spinal Cord Independence Measure (SCIM) | 12 months
  Functional improvement in SCIM after modest hypothermia

CONTACTS AND LOCATIONS:
Overall Officials: Allan D Levi, MD, PhD, Principal Investigator — University of Miami
Locations (7):
- United States (7):
  - HonorHealth Research Institute with Barrow Brain and Spine, Phoenix, Arizona
  - Jackson Memorial Hospital, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Prisma Health - University of South Carolina, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levi AD, Casella G, Green BA, Dietrich WD, Vanni S, Jagid J, Wang MY. Clinical outcomes using modest intravascular hypothermia after acute cervical spinal cord injury. Neurosurgery. 2010 Apr;66(4):670-7. doi: 10.1227/01.NEU.0000367557.77973.5F. PMID 20190669
- [Background] Dididze M, Green BA, Dietrich WD, Vanni S, Wang MY, Levi AD. Systemic hypothermia in acute cervical spinal cord injury: a case-controlled study. Spinal Cord. 2013 May;51(5):395-400. doi: 10.1038/sc.2012.161. Epub 2012 Dec 18. PMID 23247015
- [Background] Levi AD, Green BA, Wang MY, Dietrich WD, Brindle T, Vanni S, Casella G, Elhammady G, Jagid J. Clinical application of modest hypothermia after spinal cord injury. J Neurotrauma. 2009 Mar;26(3):407-15. doi: 10.1089/neu.2008.0745. PMID 19271964
- [Background] Vedantam A, Jimsheleishvili G, Harrop JS, Alberga LR, Ahmad FU, Murphy RK, Jackson JB 3rd, Rodgers RB, Levi AD. A prospective multi-center study comparing the complication profile of modest systemic hypothermia versus normothermia for acute cervical spinal cord injury. Spinal Cord. 2022 Jun;60(6):510-515. doi: 10.1038/s41393-021-00747-w. Epub 2022 Jan 10. PMID 35013548